CLINICAL TRIAL: NCT01878513
Title: Prospective Cytochrome P450 Genotyping and Clinical Outcomes in Patients With Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Jianping Zhang, Psychiatrist, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-252B
Record Dates: First submitted 2013-06-03; First posted 2013-06-17 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Psychotic Disorder Not Otherwise Specified; Severe Bipolar Disorder With Psychotic Features
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low-dose-titration condition (Experimental): Poor and intermediate CYP2D6 metabolizers will be randomized to either low-dose-titration condition or treatment-as-usual condition. In the low-dose-titration condition, patients will be treated with risperidone 0.5mg bid for 5 days, then 1mg bid for 5 days, which may be increased to 1.5mg bid for another 5 days.
  Interventions: Drug: risperidone
- Treatment-as-usual condition (Experimental): Poor and intermediate CYP2D6 metabolizers will be randomized to either low-dose-titration condition or treatment-as-usual condition. In the treatment-as-usual condition, patients will be treated with risperidone 1mg bid for 5 days, then 2mg bid for 5 days, which may be increased to 3mg bid for another 5 days.
  Interventions: Drug: risperidone
- Open-label treatment-as-usual condition (Experimental): Extensive and ultrarapid CYP2D6 metabolizers will be treated open-label in the treatment-as-usual condition. Patients will be treated with risperidone 1mg bid for 5 days, then 2mg bid for 5 days, which may be increased to 3mg bid for another 5 days.
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: risperidone — 3 levels of dosing dependent on which condition a patient is assigned to.
  Other Names: Risperdal

SUMMARY:
The aim of the study is to examine whether determining treatment strategies based upon Cytochrome P450 2D6 (CYP2D6) genotype will improve drug response rates and clinical outcome in patients with psychosis.

The investigators predict that prospectively testing CYP2D6 genotype and using this information to treat psychotic patients with risperidone will improve clinical outcomes. Specifically, CYP2D6 poor metabolizers who are treated with low dose and slow titration of risperidone will do better than those who are treated with usual dose and titration approach in terms of rates of side effects and clinical improvement.

DETAILED DESCRIPTION:
Recent large scale clinical trials have demonstrated that a substantial proportion of patients with psychotic disorders, such as schizophrenia and bipolar disorder, discontinue their antipsychotic medications due to either lack of efficacy or intolerable side effects, especially extrapyramidal symptoms (EPS). In clinical practice, it is essentially a trial and error process in deciding the best antipsychotic drug to start or switch to after a failed trial as there is little empirical data available to guide clinicians in drug selection. One promising tool, which can potentially provide valuable information to help guide medication management, is pharmacogenetic analysis of cytochrome P450 enzymes that metabolize most antipsychotics. CYP450 is a family of liver enzymes responsible for metabolizing many drugs and toxins. Genes coding for some of these enzymes have many polymorphisms, some of which produce essentially non-functional enzymes that result in poor metabolism of drugs. For example, CYP2D6 has more than 70 known mutations. Poor metabolizers may have a higher plasma concentration of a particular drug at usual dosages, which may lead to more severe side effects and potential drug discontinuation. On the other hand, rapid metabolizers tend to have a lower drug concentration in the body and may require a higher-than-usual dose to achieve clinical efficacy.

Until recently, genotyping CYP450 polymorphisms has been expensive and time-consuming, therefore clinically unfeasible. However, the recent FDA approval of a commercially available genotyping product (Roche Diagnostics, AmpliChip) as well as the greater availability of other CYP450 genotyping platforms makes it possible to quickly obtain CYP450 genotypes for clinical applications. The AmpliChip tests polymorphisms of CYP450 2D6 and 2C19, and stratifies genotype into poor metabolizer, extensive/intermediate metabolizer, and ultra-rapid metabolize groups.

Of particular importance in the treatment of psychotic disorders, such as schizophrenia and bipolar disorder with psychotic features, CYP2D6 is critical in the metabolism of risperidone, one of the most widely used atypical antipsychotic agents. Several studies have assessed CYP450 genotype in patients who were able to tolerate risperidone versus patients who were not able to. The CYP2D6 poor metabolizer phenotype was shown to be associated with risperidone side effects and discontinuation of the drug. Recent evidence suggest that intermediate metabolizers also tend to have higher rates of side effects when taking regular doses of risperidone.

A major limitation of the previous studies is their case-control and retrospective design. To date, no study has prospectively examined the clinical utility of CYP450 polymorphism genotyping in psychosis. Therefore, we will conduct a prospective study in which patients with psychosis undergo CYP450 genotyping at study entry, and antipsychotic drug dosage is determined by CYP2D6 genotype.

In this study, we are conducting a randomized double blind trial of risperidone treatment for psychotic patients who are admitted to inpatient units due to acute relapse. We anticipate to recruit 264 subjects and test their CYP2D6 polymorphism genotypes, based on which they will be randomly assigned to either a low dose slow titration group or a treatment as usual group. They will be assessed every five days for 15 days, and then at follow-ups at 4-weeks and 6-weeks from study entry.

It is hoped that this study will provide prospective data on whether pharmacogenetic information such as CYP450 2D6 polymorphism genotypes can have a significant clinical impact on patients with psychotic disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60;
2. DSM-IV(Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition) diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, or psychotic disorder NOS (Not otherwise specified), bipolar disorder with psychotic features
3. Having moderate to severe psychotic symptoms resulting in inpatient admission
4. Able to provide informed consent

Exclusion Criteria:

1. Evidence of serious medical conditions,
2. Evidence of liver disease, as shown in elevated liver function test
3. Female patients who are pregnant or breast feeding;
4. History of allergic reactions to risperidone or Invega;
5. History of risperidone or Invega treatment failure.
6. History of receiving any long-acting injectable form of antipsychotic medications such as haloperidol decanoate, fluphenazine decanoate, Risperdal Consta, Invega Sustenna, and Zyprexa IntraMuscular in the past two months.
7. History of treatment with clozapine.
8. Medications that potentially interfere with the CYP450 2D9 enzyme family, including bupropion, fluoxetine, paroxetine, duloxetine, sertraline, cinacalcet, quinidine, terbinafine, amiodarone, and cimetidine, and as per clinical review by study physicians.
9. Patients who are not able to provide informed consent due to impairment in decision-making capacity.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2009-09-23 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Efficacy | 6 weeks or discharge up to 6 weeks
  Scores on:
  1. Schedule for Assessment of Negative Symptoms (SANS)
  2. Brief Psychiatric Rating Scale (BPRS)
  3. Global Impression - Improvement scale (CGI-I)

SECONDARY OUTCOMES:
Adverse Drug Effects | 6 weeks, discharge or discontinuation up to 6 weeks
  As measured by:
  1. Hillside Hospital Adverse Events Rating Scale
  2. Abnormal Involuntary Movement Scale (AIMS)
  3. Barnes Rating Scale for Drug-Induced Akathisia
  4. Simpson-Angus Rating Scale for Extrapyramidal symptoms

OTHER OUTCOMES:
Number of days before discontinuation | 6 weeks, discontinuation or discharge up to 6 weeks
Days of Inpatient Stay | 6 weeks, discontinuation or discharge up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Zhang, MD, PhD, Principal Investigator — Zucker Hillside Hospital, Division of Psychiatry Research
Locations (1):
- Zucker Hillside Hospital, Glen Oaks, New York, United States

IPD SHARING:
Plan to Share IPD: No